CLINICAL TRIAL: NCT02702739
Title: Efficacy and Safety of Sofosbuvir/Simeprevir Plus a Flat Dose of Ribavirin in Genotype 1 Elderly Cirrhotic Patients: a Real Life Study
Brief Title: Sofosbuvir/Simeprevir Plus a Flat Dose of Ribavirin in Genotype 1 Elderly HCV Cirrhotic Patients
Acronym: HCV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliera San Camillo Forlanini (Other)
Responsible Party: Principal Investigator, Adriano Pellicelli, Director Liver Unit, Azienda Ospedaliera San Camillo Forlanini
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDAAA 801
Record Dates: First submitted 2016-02-23; First posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Sofosbuvir; Simeprevir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (<65 years) (Active Comparator): Group I treated with Sofosbuvir 400mg/day/Simeprevir 150mg/day /Ribavirin 800mg/day for 12 weeks
  Interventions: Drug: Sofosbuvir 400mg/day/Simeprevir 150mg/day /Ribavirin 800mg/day for 12 weeks
- Group II (>65 years) (Active Comparator): Group II treated with Sofosbuvir 400mg/day/Simeprevir 150mg/day /Ribavirin 800mg/day for 12 weeks
  Interventions: Drug: Sofosbuvir 400mg/day/Simeprevir 150mg/day /Ribavirin 800mg/day for 12 weeks

INTERVENTIONS:
Drug: Sofosbuvir 400mg/day/Simeprevir 150mg/day /Ribavirin 800mg/day for 12 weeks — Sofosbuvir 400 mg/day/Simeprevir 150 mg/day /Ribavirin 800/day for 12 weeks
  Other Names: Sovaldi Olysio Copegus

SUMMARY:
The proportion of HCV infected patients over age 65 years in Western countries is increasing. This growth and the advent of new antiviral therapy bring into the question the real world efficacy and safety of the combination of Sofosbuvir and Simeprevir (SOF/SMV) plus a flat dose of ribavirin (RBV) in elderly patients compared to younger patients.

DETAILED DESCRIPTION:
The proportion of HCV infected patients over age 65 years in Western countries is increasing. This growth and the advent of new antiviral therapy bring into the question the real world efficacy and safety of the combination of Sofosbuvir and Simeprevir (SOF/SMV) plus a flat dose of ribavirin (RBV) in elderly patients (Group II) compared to younger patients (Group I) Multicenter, real world investigation study of once daily treatment with SOF 400 mg + SMV 150 mg with a flat dose of RBV 800 mg/day for a duration of 12 weeks in treatment naïve or experienced HCV genotype 1-infected patients with compensated cirrhosis.To evaluate efficacy, tollerability and safety of SOF/SMV/RBV in two different Group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Naive or experienced patients with genotype 1 compensated cirrhosis

Exclusion Criteria:

* HIV and hepatitis B infection, active hepatocellular carcinoma (HCC), decompensated cirrhosis, history of organ transplant, severe psychiatric disorders or treatment with drugs that showed an interaction with antiviral treatment.

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Sustained virological response week 12 after the end of treatment | up 12 weeks
  to evaluate the efficacy in term of sustained virological response after 12 weeks from the end of treatment in the two Groups of patients

SECONDARY OUTCOMES:
Adverse events and severe adverse events during the treatment period | up 12 weeks
  To report Adverse events and severe adverse events during the treatment period in the two Groups of patients

CONTACTS AND LOCATIONS:
Overall Officials: Adriano M Pellicelli, MD, Study Director — AO San Camillo Forlanini ROme ITALY
Locations (1):
- AO San Camillo Forlanini, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pellicelli AM, Romano M, Guarascio P, Vignally P. Which is the real efficacy of pegylated interferon alpha 2a or 2b plus ribavirin in HCV infected patients with advanced fibrosis? J Hepatol. 2012 Sep;57(3):704-5. doi: 10.1016/j.jhep.2012.03.008. Epub 2012 Apr 14. No abstract available. PMID 22510262
- [Result] Fontana RJ, Brown RS Jr, Moreno-Zamora A, Prieto M, Joshi S, Londono MC, Herzer K, Chacko KR, Stauber RE, Knop V, Jafri SM, Castells L, Ferenci P, Torti C, Durand CM, Loiacono L, Lionetti R, Bahirwani R, Weiland O, Mubarak A, ElSharkawy AM, Stadler B, Montalbano M, Berg C, Pellicelli AM, Stenmark S, Vekeman F, Ionescu-Ittu R, Emond B, Reddy KR. Daclatasvir combined with sofosbuvir or simeprevir in liver transplant recipients with severe recurrent hepatitis C infection. Liver Transpl. 2016 Apr;22(4):446-58. doi: 10.1002/lt.24416. PMID 26890629
- [Result] Pellicelli AM, Montalbano M, Lionetti R, Durand C, Ferenci P, D'Offizi G, Knop V, Telese A, Lenci I, Andreoli A, Zeuzem S, Angelico M. Sofosbuvir plus daclatasvir for post-transplant recurrent hepatitis C: potent antiviral activity but no clinical benefit if treatment is given late. Dig Liver Dis. 2014 Oct;46(10):923-7. doi: 10.1016/j.dld.2014.06.004. Epub 2014 Jul 3. PMID 24997638
- [Derived] Pellicelli AM, Pace Palitti V, Vignally P, Ceccherini-Silberstein F, Siciliano M, Giannelli V, Moretti A, Tarquini P, Scifo G, Messina V, Ascione A, Izzi A, Marignani M, D'Ambrosio C, Fondacaro L, Ettorre GM, Ialongo P, Sacco R, Perno CF, Barbarini G; CLEO Group. Efficacy and safety of sofosbuvir/simeprevir plus flat dose ribavirin in genotype 1 elderly cirrhotic patients: A real-life study. Liver Int. 2017 May;37(5):653-661. doi: 10.1111/liv.13288. Epub 2016 Dec 15. PMID 27782373